CLINICAL TRIAL: NCT03697083
Title: Reminders Through Association & Prescription Adherence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The primary hypotheses were unsupported with half of the data collected.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 825556
Record Dates: First submitted 2018-08-28; First posted 2018-10-05 (Actual); Results first posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-06

CONDITIONS: Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reminders Through Association Arm (Experimental): participants will be prompted to think of a reminder cue that will help them remember to pick up the prescription.
  Interventions: Other: Reminders Through Association
- Active Control Arm (Active Comparator): Participants will be asked to think about where they will store their prescription.
  Interventions: Other: Active Control
- Baseline Control Arm (Active Comparator): Participants are thanked for enrolling in the reminder program.
  Interventions: Other: Baseline Control

INTERVENTIONS:
Other: Reminders Through Association — Participants receive 8 text messages asking them to think of a reminder cue that will help them remember to pick up the prescription and use the cue.
  Arms: Reminders Through Association Arm
Other: Active Control — Participants receive 8 text messages asking them to think of where they plan to store their medication once they pick it up and to think about that location on their intended date of pickup.
  Arms: Active Control Arm
Other: Baseline Control — Participants receive 1 text message thanking participants for enrolling in the reminder program. Participants are not contacted further.
  Arms: Baseline Control Arm

SUMMARY:
The purpose of this study is to develop behavioral interventions that provide effective tools that policy makers can use to help individuals avoid forgetting to follow-through on important behaviors and for individuals to use to help themselves. In the investigators past research, they have shown that reminders through association work in the lab setting. The investigators seek to understand how this strategy can work in the field, especially when people are trying to fulfill a health outcome.

DETAILED DESCRIPTION:
Participants enter an online survey where they are asked to confirm that they plan to pick up a prescription, state what day they plan to pick up their prescription, and indicate the type of location where the prescription will be picked up (e.g., pharmacy, hospital, doctors office, etc.). Participants are asked to participate in a prescription reminder program in which they will receive up to eight text messages from the researchers and send up to three text messages to the researchers. Participants are then quizzed about the reminder program to ensure they understand what they are signing up for. Participants are further told that if they follow the directions outlined in the program they will be compensated for participating in this survey via their phone number.

Participants who wish to enroll in the reminder program will initiate the text messaging by texting "STARTXXXX" to number provided. This validates that the participants received the message, have the capacity to text, and are willing to text. Participants are then randomly assigned to one of three conditions. In the treatment condition, participants will be prompted to think of a reminder cue that will help them remember to pick up the prescription. In the active control condition, participants will be asked to think about where they will store their prescription. Participants in the baseline control condition will simply be thanked for enrolling.

Participants in the treatment and active control conditions then receive a series of text messages prior to the scheduled pick up date reminding them to pick up their medication. In addition, the text message will prompt participants to text a picture of their prescription receipt to validate that they followed-through on their behavior. If participants text us a picture of their receipt that follows the guidelines outlined in the survey, participants are compensated.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be capable of sending and receiving text and picture messages on their phone.

Exclusion Criteria:

* Participants will only be excluded if they participated in the pilot study in which the investigators enrolled 150 participants. These participants will be excluded when they attempt to text the investigators to enroll.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 777 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Milkman, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reminders Through Association Arm | Active Control Arm | Baseline Control Arm
Started | 262 | 260 | 255
Completed | 262 | 250 | 255
Not Completed | 0 | 10 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reminders Through Association Arm | Active Control Arm | Baseline Control Arm | Total
Number analyzed (Participants) | 262 | 260 | 255 | 777
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (13.6) | 41.2 (13.8) | 40.44 (13.4) | 41 (13.58)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 39 | 35 | 45 | 119
  Female | 218 | 218 | 205 | 641
  Other | 4 | 6 | 4 | 14
  Prefer not to specify | 1 | 1 | 1 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Picking up Prescription on Intended Date of Pickup
Description: At the beginning of the study, participants indicate the date they plan to pick up their prescription. Participants are later asked to text a picture of their prescription receipt to the experimenter after they complete the prescription reminder program. The receipt must satisfy three criteria:
  1. The receipt must show that a prescription was purchased.
  2. The receipt must show the date of purchase. This date of purchase must match the participant's intended pick up date.
  3. The participant must write the word "End" on their receipt. Upon receiving the picture text, one research assistant will verify that the image of the receipt satisfies all three criteria.
  the investigators' primary dependent variable is binary taking the value one if the participant sends a picture of their receipt to the investigators that satisfies all criteria stated above and taking the value zero if otherwise.
Time Frame: The time frame can range from less than 1 day to a maximum of 7 days.
Measure: Mean (Standard Deviation); unit: percentage of prescriptions pickuped
Arm/Group | Reminders Through Association Arm | Active Control Arm | Baseline Control Arm
Number analyzed (Participants) | 262 | 260 | 255
percentage of prescriptions pickuped | 46 (.50) | 46 (.50) | 15 (.36)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during data collection and one week after recruitment ended.
Description: This intervention was solely to help people pick up their prescriptions. Participants only received a series of text messages so there was not risk serious adverse events.
Arm/Group | Reminders Through Association Arm | Active Control Arm | Baseline Control Arm
All-Cause Mortality (participants affected / at risk) | 0/262 | 0/260 | 0/255
Serious Adverse Events (participants affected / at risk) | 0/262 | 0/260 | 0/255
Other Adverse Events (participants affected / at risk) | 0/262 | 0/260 | 0/255

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT03697083/Prot_SAP_000.pdf